CLINICAL TRIAL: NCT05071248
Title: Evaluation of the Effect of Robot-assisted Early Mobilization on Critically Ill Patients, on the Mobilisation Behaviour and Experience of Mobilizing Professionals and Organisational Processes in an Intensive Care Unit
Brief Title: Evaluation of the Effect of Robot-assisted Early Mobilization - Project MobiStaR
Acronym: MobiStaR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government); Catholic University of Eichstätt-Ingolstadt (Other)
Responsible Party: Principal Investigator, Dr. Uli Fischer, Head of executive department nursing science, Ludwig-Maximilians - University of Munich
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: 16SV842
Record Dates: First submitted 2021-08-27; First posted 2021-10-08 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: Patient Activation; Mobilization; Robotics
Keywords: robotics; intensive care unit; VEM; very early mobilization; feasibility; effects on patients' outcomes; mobilising professionals; Sonography; mixed methods; routine data; observations; interview; nursing sciences; physiotherapy; nurse
MeSH Terms: conditions — Patient Participation

STUDY DESIGN:
Intervention Model Description: The present study is a monocentric, prospective intervention study designed to evaluate the feasibility and
  * to evaluate the feasibility and integration in the setting of the intensive care unit.
  * the behavior and experience of the mobilizing specialists of the robot-assisted VEM is to be evaluated longitudinally (three data collection points).
  * to compare robot-assisted VEM in critically ill ICU patients with non-robot-assisted early mobilization according to the standard of care of a historical patient population.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patients with robot-assisted early mobilization (Active Comparator): All patients will receive a physical examination at various time points to assess physical functionality and muscle strength, as well as a sonographic examination of leg muscles, diaphragm, and lungs. These examinations should be performed on day -1 (preoperatively), on postoperative days 1,2,3, then once a week if the patient remains in the ICU, on day 28, on the day of discharge from the ICU, and on a follow-up examination approximately 3 months after discharge from the ICU.The follow-up examination should only take place if the patients present themselves at the hospital anyway due to medically indicated follow-up examinations (not study-related). Alternatively, patients can be asked about their condition by telephone.
  Interventions: Device: VEMO (Reactive Robotics GmbH)
- patients with conventional early mobilization (historic group) (No Intervention): All patients fulfill the same criteria like the intervention group and receive conventional early mobilization.

INTERVENTIONS:
Device: VEMO (Reactive Robotics GmbH) — The robot used for early mobilization is able to verticalize the patients in their bed without transfer and to generate a movement of the legs that measures and supports the patients' own movement. The device meets the requirements for mobilizing critically ill patients in an intensive care unit, maintaining hygiene standards and providing the best possible support for the patient's own movement.
  Arms: patients with robot-assisted early mobilization

SUMMARY:
Within the MobiStaR project the adaptation of procedures in an intensive care unit combined with the use of this robotic system will create the conditions to increase the mobilization rate of critically ill intensive care patients significantly, possibly thereby increasing the rehabilitation outcomes for these patients and developing a new standard of care for robot-assisted early mobilization.

The intervention study will assess the organizational feasibility of robot-assisted early mobilization (starting in the first 72 hours after admission to the ICU), the behavior and experience of the mobilizing professionals and the effects on patient outcomes in terms of ventilation time, muscle mass (sonographic examination) and physical activity (measured by established scores such as Functional Status Score for ICU (FSS-ICU) and Medical Research Council (MRC) classification).

DETAILED DESCRIPTION:
Early mobilization means the mobilization of critically ill patients in the early course after admission to the intensive care unit. The positive influence of early mobilization of critically ill patients on various aspects of patient outcomes has already been demonstrated. However, the implementation of early mobilization in clinical practice is difficult. Especially the high personnel effort is a barrier.

The Munich-based company Reactive Robotics (RR) is currently developing the world's first adaptive robotic assistance system VEMO©, which has CE approval for the planned indication and is to be used in the medium term for mobilizing intensive care patients.

Within the MobiStaR project, the adaptation of procedures in an intensive care unit combined with the use of this robotic system will create the conditions to significantly increase the mobilization rate of critically ill intensive care patients, possibly thereby increasing the rehabilitation results for these patients and developing a new standard of care for robot-assisted early mobilization. In this project, the robotic system will be used in anesthesiology intensive care units of the Ludwigs-Maximilians-University hospital.

Within this study, the effects of robot-assisted early mobilization will now be evaluated. This study comprises three study arms, in which (1) the feasibility and practicability of robot-assisted early mobilization, (2) the behavior and experience of the mobilizing professionals, and (3) the effect on patient outcomes will be evaluated.

The study is monocentric, prospective, interventional, does not include invasive procedures or blood sampling and has multiple data collection time points.

1. The feasibility of robot-assisted early mobilization surveys concomitantly how many VEM therapies can be implemented in how many patients as well as if and which adverse events occur.
2. The behavior and experience of the mobilizing professionals will be evaluated by using episodic interviews and standardized observations. Nurses with advanced training in anesthesia and intensive care, nurses and physiotherapists who have at least three years of professional experience in an intensive care unit as well as medical specialists with completed specialist training or a leading position in the intensive care unit will be included.
3. The effects on patient outcomes, primarily ventilation duration, muscle mass (sonographic examination) and physical activity (measured by established scores such as FSS-ICU and MRC classification), will be measured at different time points and compared with a historical patient population. Secondary factors such as delirium incidence, hemodynamic parameters, respiratory parameters but also longitudinal parameters such as ICU and hospital length of stay will be analyzed from routine data/patient records. Informed consenting patients undergoing a planned surgical procedure that is postoperatively associated with intensive care treatment and an anticipated duration of ventilation of more than 48 hours will be included. These patients will receive standardized early mobilization using the robotic system at either ten frequencies or for seven days. No invasive procedures such as blood sampling will be performed as part of the study. Outcomes will be compared with a historical comparison group to evaluate the effect of robot-assisted VEM (very early mobilization). Approximately 30 patients will be included. The outcomes will be compared with those of a historical group (n=30) treated with conventional early mobilization.

The intervention is planned for a duration of five to six months starting in September 2021.

ELIGIBILITY:
Inclusion Criteria:

* planned surgical intervention
* postoperative intensive medical and therapeutic treatment
* expected duration of ventilation > 48 hours
* age ≥ 18 years
* preoperative informed consent by the patients in the study
* weight >45 kg and <135 kg
* body height >1.50 m and <1.95 m

Exclusion Criteria:

* patient refusal to participate in the study
* unable to give consent
* chronically bedridden before inclusion
* clinical Frailty Scale ≥ 7
* chronic ventilation (over 24h) before ICU admission
* increased intracranial pressure / risk for increased intracranial pressure / recent cerebral hemorrhage
* pregnancy
* pre-existing neuromuscular disease resulting in chronic limitation of strength and efficiency
* sternotomy / sternectomy during surgical procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2022-04-15 (Actual); Study Completion 2022-05-15 (Actual)

PRIMARY OUTCOMES:
Evaluation of the effect of robot-assisted early mobilization on critically ill patients - Ventilation duration | 6 months
  changes in ventilation duration (in hours) in comparison to a historical patient group
Evaluation of the effect of robot-assisted early mobilization on critically ill patients - sonographic examination Area of the M.rec.femoris | 6 months
  muscle mass (sonographic examination, in millimeters): Area of the M. rec. femoris in comparison to a historical patient group (in cm²)
Evaluation of the effect of robot-assisted early mobilization on critically ill patients - sonographic examination thickness M. quad. femoris | 6 months
  muscle mass: Thickness M. quad. Femoris (in cm²) in comparison to a historical patient group
Evaluation of the effect of robot-assisted early mobilization on critically ill patients - sonographic examination- motility diaphragm breathing | 6 months
  muscle mass: motility of the diaphragm during breathing (in cm) in comparison to a historical patient group
Evaluation of the effect of robot-assisted early mobilization on critically ill patients - sonographic examination thickness diaphragm inspiration | 6 months
  muscle mass: Thickness of diaphragm during inspiration (in cm) in comparison to a historical patient group
Evaluation of the effect of robot-assisted early mobilization on critically ill patients - sonographic examination thickness diaphragm exhalation | 6 months
  muscle mass: Thickness of diaphragm during exhalation (in cm) in comparison to a historical patient group
Evaluation of the effect of robot-assisted early mobilization on critically ill patients - physical activity - FSS-ICU | 6 months
  physical activity measured using the score FSS-ICU (0 -35) in comparison to a historical patient group. A higher value means a better outcome.
Evaluation of the effect of robot-assisted early mobilization on critically ill patients - physical activity | 6 months
  physical activity on upper and lower extremity measured using the Medical Research Council (MRC) score in comparison to a historical patient group. (0=absent muscle contraction, 1=visible muscle contraction, 2=movement when gravity is eliminated, 3=active movement against gravity, 4=active movement against resistance, 5=normal strength.)
Behavior and experience of the mobilizing professionals - qualitative interviews | 6 months
  subjectively experienced emotions, motivating and challenging factors - evaluated with a semi-structured interview guideline
Behavior and experience of the mobilizing professionals - qualitative observations | 6 months
  behavior and body posture during the mobilization - evaluated with a standardized observation sheet
Feasibility in organizational processes - eligible patients | 6 months
  Frequency of eligible patients (count per week: included patients in the study/ new eligible patients in the ICUs)
Feasibility in organizational processes - mobilizations | 6 months
  frequency of robot-assisted mobilizations (per patient per day)
Feasibility in organizational processes - adverse events | 6 months
  adverse events (count of patient-related, user-related or technology-related adverse events)

SECONDARY OUTCOMES:
Delir | 6 months
  Delir incidence using the CAM ICU: number of days without Delir. 1 = pathological; 2 = normal; 3 = not performed in comparison to a historical patient group
Consciousness | 6 months
  level of consciousness using the Glasgow Coma Scale (3-15) in comparison to a historical patient group
Sedation level | 6 months
  Sedation level using the Richmond Agitation Sedation Scale (RASS) (-5 - +5) in comparison to a historical patient group
Pain (VAS) | 6 months
  Pain - with the use of the Visual Analog Scale (VAS) (before and after mobilization) (0-10) in comparison to a historical patient group
health related quality of life | 6 months
  Health-related quality of life after 3 months using the the SF-36 (Short form questionnaire) (0-100) in comparison to a historical patient group
Blood pressure | 6 months
  hemodynamics - Blood pressure (in mmHg) in comparison to a historical patient group
catecholamine demand | 6 months
  hemodynamics - catecholamine demand (cumulative over 24 hours) in comparison to a historical patient group
heart rate | 6 months
  hemodynamics - heart rate (1/min) in comparison to a historical patient group
cardiac output | 6 months
  hemodynamics - Cardiac output (in l/min) in comparison to a historical patient group
oxygen consumption | 6 months
  hemodynamics - Oxygen consumption (in l) in comparison to a historical patient group
respiration | 6 months
  respiration- Maximum respiratory rate for 24h in comparison to a historical patient group
ICU Score - SOFA | 6 months
  ICU Scores like Sepsis-related organ failure assessment score (SOFA) (0-24) in comparison to a historical patient group. A higher value means a worse outcome.
ICU Scores - APACHE II | 6 months
  ICU Scores like Acute Physiology and Chronic Health Disease Classification System II (APACHE II) (0-71) in comparison to a historical patient group. A higher value means a worse outcome.
ICU Scores - SAPS II | 6 months
  ICU Scores like Simplified Acute Physiology Score II (SAPS II) (0-163) in comparison to a historical patient group. A higher value means a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Zoller, PD Dr., Principal Investigator — Ludwig-Maximilians - University of Munich; Inge Eberl, Prof. Dr., Principal Investigator — Catholic University of Eichstätt-Ingolstadt; Eduard Kraft, PD Dr., Principal Investigator — Ludwig-Maximilians - University of Munich; Uli Fischer, Dr., Principal Investigator — Ludwig-Maximilians - University of Munich
Locations (1):
- LudwigMaximilians, Munich, Bavaria, Germany

REFERENCES:
- [Derived] Huebner L, Warmbein A, Scharf C, Schroeder I, Manz K, Rathgeber I, Gutmann M, Biebl J, Mehler-Klamt A, Huber J, Eberl I, Kraft E, Fischer U, Zoller M. Effects of robotic-assisted early mobilization versus conventional mobilization in intensive care unit patients: prospective interventional cohort study with retrospective control group analysis. Crit Care. 2024 Apr 6;28(1):112. doi: 10.1186/s13054-024-04896-1. PMID 38582934
- [Derived] Warmbein A, Hubner L, Rathgeber I, Mehler-Klamt AC, Huber J, Schroeder I, Scharf C, Gutmann M, Biebl J, Manz K, Kraft E, Eberl I, Zoller M, Fischer U. Robot-assisted early mobilization for intensive care unit patients: Feasibility and first-time clinical use. Int J Nurs Stud. 2024 Apr;152:104702. doi: 10.1016/j.ijnurstu.2024.104702. Epub 2024 Jan 26. PMID 38350342
- [Derived] Warmbein A, Schroeder I, Mehler-Klamt A, Rathgeber I, Huber J, Scharf C, Hubner L, Gutmann M, Biebl J, Lorenz A, Kraft E, Zoller M, Eberl I, Fischer U. Robot-assisted early mobilization of intensive care patients: a feasibility study protocol. Pilot Feasibility Stud. 2022 Nov 5;8(1):236. doi: 10.1186/s40814-022-01191-0. PMID 36333746

DOCUMENTS (1):
  • Study Protocol (2021-05-27): https://cdn.clinicaltrials.gov/large-docs/48/NCT05071248/Prot_000.pdf